CLINICAL TRIAL: NCT00577499
Title: Effect of Lubiprostone on Nutritional Status and Pulmonary Function in Adults With Cystic Fibrosis
Status: Terminated | Type: Observational
Why Stopped: Recruitment was suboptimal
Sponsor: University of Arkansas (Other)
Collaborators: American Society of Health-System Pharmacists Research and Education Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 84063; 07-JI-166
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Cystic Fibrosis; Constipation; Nutrition
Keywords: cystic fibrosis; constipation; lubiprostone; nutrition; pulmonary function
MeSH Terms: conditions — Cystic Fibrosis; Constipation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Only group: adult cystic fibrosis patients who are not at goal body mass index and have started lubiprostone therapy within one month of study enrollment

SUMMARY:
Cystic fibrosis (CF) results in thickened secretions in multiple organ systems including the lungs and gastrointestinal (GI) tract. Patients commonly suffer from nutritional deficiency, and achieving and maintaining adequate nutrition is an important goal of therapy because it is positively correlated with lung function. Lubiprostone activates chloride channels in the GI tract. Because its mechanism of action closely parallels the disease pathology, lubiprostone has the potential to provide GI benefits beyond the relief of constipation. This project is an observational study to examine the effects of lubiprostone on nutritional status and lung function in adults with CF. Our hypothesis is that lubiprostone will have beneficial effects on nutritional status.

DETAILED DESCRIPTION:
Background: Cystic fibrosis (CF) affects an estimated 30,000 people in the United States. It is caused by a mutation in the gene encoding a protein called cystic fibrosis transmembrane regulator (CFTR). This protein functions as a chloride channel in epithelial cells of multiple organ systems. The mutation results in a dysfunctional or absent CFTR channel and a decrease in chloride secretion, which results in thickened secretions in multiple organ systems including the lungs and gastrointestinal (GI) tract. This patient population commonly suffers from nutritional deficiency, and achieving and maintaining normal nutritional status is an important goal of therapy as body mass index (BMI) is positively correlated with forced expiratory volume in 1 second (FEV1), a measure of pulmonary function. Lubiprostone activates type 2 chloride channels (ClC-2) on the apical membrane of GI epithelial cells. Because its mechanism of action closely parallels the disease pathology, lubiprostone has the potential to provide GI benefits beyond the relief of constipation. Objectives: The proposed pilot project is a prospective observational study to examine the effects of lubiprostone in adults with CF. The specific aims are to determine the effects of lubiprostone on: 1) nutritional markers and 2) pulmonary function in adults with CF. Methods: Adults with CF who are currently taking lubiprostone chronically will be sought for enrollment. Study subjects will be followed for approximately 3-months with serial assessment of indicators of nutrition and pulmonary function. Nutritional markers to be measured include body weight, albumin, prealbumin, and vitamins A, D, and E. Pulmonary function will be assessed by pulmonary function tests, a survey to monitor for symptoms of pulmonary exacerbation, and monitoring of the frequency of hospitalizations and IV antibiotic use. Expected Results: We expect to see a beneficial effect on nutritional markers, body weight, and BMI. We hope this translates into a concomitant improvement in pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

* Planning or currently on chronic lubiprostone therapy (chronic is defined as at least one 24 microgram capsule by mouth every other day
* Body mass index (BMI) of less than 22 for females and less than 23 for males at the initiation of chronic lubiprostone therapy
* Initiation of chronic lubiprostone therapy within 1 month of enrollment
* Age over 18
* Currently taking a multivitamin

Exclusion Criteria:

* History of noncompliance with medications and other CF therapies
* History of hospital admissions for CF exacerbations of ≥2 in the last 6 months
* FEV1 les than 40% of expected (severe dysfunction) at most recent assessment in the ambulatory setting
* Currently registered on a lung transplant waiting list
* Any other condition, in the opinion of the investigators, that interferes with the ability of the study subject to comply with study requirements, confers significant risk, or limits the ability of the subject to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult cystic fibrosis clinic
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2007-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
body mass index | 3 months

SECONDARY OUTCOMES:
pulmonary function tests | 3 months
cystic fibrosis clinical score | 3 months
Serum nutritional markers (vitamins A, D, E; albumin; prealbumin) | 3 months
24-hour diet recall | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine O'Brien, PharmD, Principal Investigator — University of Arkansas